CLINICAL TRIAL: NCT00962065
Title: A Phase 2, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Determine the Safety and Efficacy of Orally Administered LX4211 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study of LX4211 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Joel P. Freiman, MD, MPH - Medical Director, Lexicon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LX4211.1-201-DM; LX4211.201
Record Dates: First submitted 2009-08-10; First posted 2009-08-19 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Experimental): A low dose of LX4211; daily oral intake for 28 days
  Interventions: Drug: LX4211 Low Dose
- High Dose (Experimental): A high dose of LX4211; daily oral intake for 28 days
  Interventions: Drug: LX4211 High Dose
- Placebo (Placebo Comparator): Matching placebo dosing with daily oral intake for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LX4211 Low Dose — A low dose of LX4211; daily oral intake for 28 days
  Arms: Low Dose
Drug: LX4211 High Dose — A high dose of LX4211; daily oral intake for 28 days
  Arms: High Dose
Drug: Placebo — Matching placebo dosing with daily oral intake for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of LX4211 versus a placebo control in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (non-childbearing potential), aged 18-65 years
* Diagnosis of Type 2 diabetes mellitus for at least 6 months prior to screening
* Fasting plasma glucose ≤ 240 mg/dL prior to metformin washout
* Body mass index < 42 kg/m^2
* HbA1c value of 7 to 11%
* C-peptide ≥ 1.0 ng/mL
* Ability to provide written informed consent

Exclusion Criteria:

* History of Type 1 diabetes mellitus, diabetic ketoacidosis, hyperosmolar nonketotic syndrome, incontinence, or nocturia
* Use of any blood glucose lowering agent other than metformin
* Prior exposure to insulin, thiazide, or loop diuretics within 4 weeks prior to screening
* Laboratory or electrocardiogram abnormalities deemed significant by the Sponsor or the Investigator
* Positive test result for glutamic acid decarboxylase (GAD) antibody
* Surgery within 6 months of screening
* Exposure to any investigational agent or participation in any investigational trial within 30 days prior to Day 1
* Hypersensitivity to an SGLT2 inhibitor
* History of drug or alcohol abuse within the last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel P. Freiman, MD, MPH, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Zambrowicz B, Freiman J, Brown PM, Frazier KS, Turnage A, Bronner J, Ruff D, Shadoan M, Banks P, Mseeh F, Rawlins DB, Goodwin NC, Mabon R, Harrison BA, Wilson A, Sands A, Powell DR. LX4211, a dual SGLT1/SGLT2 inhibitor, improved glycemic control in patients with type 2 diabetes in a randomized, placebo-controlled trial. Clin Pharmacol Ther. 2012 Aug;92(2):158-69. doi: 10.1038/clpt.2012.58. Epub 2012 Jul 4. PMID 22739142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center trial in the United States, with 1 investigator participating.
Pre-assignment Details: There was a 14-day washout period and a 5-day diet stabilization period prior to randomization.
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (6.07) | 52.3 (8.40) | 54.5 (7.23) | 53.2 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 6 | 16
  Male | 6 | 8 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 11 | 29
  Not Hispanic or Latino | 4 | 2 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Black or African American | 2 | 0 | 0 | 2
  White or Caucasian | 10 | 10 | 12 | 32
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Day 28 in 24-hour Urinary Glucose Excretion
Description: To assess 24-hour urinary glucose excretion, urine was collected over a 24-hour period and evaluated for glucose concentration.
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12
grams | 35.729 [26.207 to 45.252] | 47.085 [37.562 to 56.608] | -0.965 [-10.768 to 8.838]

2. Secondary Outcome: Change From Baseline at Day 29 in Fasting Plasma Glucose
Time Frame: Baseline to Day 29
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12
mg/dL | -52.3 [-67.7 to -36.9] | -67.8 [-83.2 to -52.4] | -12.3 [-28.0 to 3.4]

3. Secondary Outcome: Change From Baseline at Day 28 in Plasma HbA1c
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Percent | -1.15 [-1.58 to -0.72] | -1.25 [-1.68 to -0.82] | -0.49 [-0.93 to -0.05]

4. Secondary Outcome: Change From Baseline at Day 28 in Plasma Fructosamine Level
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: µmol/L
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12
µmol/L | -24.5 [-39.5 to -9.5] | -24.9 [-39.9 to -9.9] | 18.1 [2.7 to 33.5]

5. Secondary Outcome: Change From Baseline at Day 28 in Mean Arterial Pressure
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12
mm Hg
  Standing | -8.6 [-13.8 to -3.4] | -5.6 [-10.8 to -0.4] | -3.8 [-9.2 to 1.6]
  Seated | -7.3 [-12.3 to -2.4] | -7.9 [-12.9 to -3.0] | -3.4 [-8.5 to 1.8]
  Supine | -8.2 [-13.2 to -3.3] | -6.1 [-11.0 to -1.2] | -4.9 [-10.1 to 0.2]

6. Secondary Outcome: Change From Baseline at Day 28 in Triglycerides
Time Frame: Baseline to Day 28
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 12 | 12
mg/dL | -66.6 [-105.2 to -28.0] | -62.8 [-101.3 to -24.2] | -20.2 [-60.5 to 20.1]

ADVERSE EVENTS:
Time Frame: Adverse events were followed during the treatment period.
Arm/Group | Low Dose | High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/12 | 8/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=12) | High Dose (N=12) | Placebo (N=12)
Headache (Nervous system disorders) | 5 (10) | 1 (15) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (14) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Pyuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteriuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritis genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires that written permission be given before the PI can release any data publicly.